CLINICAL TRIAL: NCT07093619
Title: Evaluating the Utility of Implementing Microfluids for Sperm Preparation Compared to Conventional Method of Density Gradient Centrifugation in a PGT-A Program: a Sibling Oocyte Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Andrea Abdala, Senior Clinical Embryologist, ART Fertility Clinics LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2504-ABU-011-AAb
Record Dates: First submitted 2025-06-27; First posted 2025-07-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Semen Analysis; ICSI; PGT-A
Keywords: IVF; Sperm Preparation; euploid; fertilization rate; blastulation rate; morphokinetics

STUDY DESIGN:
Intervention Model Description: 50% microfluids group and 50% gradient group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperm Source obtained by microfluids (Other)
  Interventions: Device: FERTILE Plus
- Sperm Source obtained by gradients (Other)
  Interventions: Device: FERTILE Plus

INTERVENTIONS:
Device: FERTILE Plus — The FERTILE PLUS™ method is a standardized method with an easy-to-follow protocol that is far less dependent on the skill or experience of the embryologist than other methods, such as density gradients. The FERTILE PLUS™ (850 µL) Sperm Sorting Chip is a single-use, flow-free, dual chambered, microfluidic-based sperm sorting device. FERTILE PLUS™ was previously known as Zymot, prior to a name change by the manufacturer. The lower chamber contains a sample inlet and fluid channel separated from the upper collection chamber by a microporous membrane with 8-μm pores, demonstrated as the optimal size for selection of sperm with higher motility and normal morphology [18].

SUMMARY:
In assisted reproductive technology (ART), sperm preparation aims to select the most viable sperm for ICSI. Unlike conventional methods like density gradients or sperm washing, microfluidic techniques mimic natural selection in the female reproductive tract by using laminar flow without centrifugation, reducing the risk of DNA damage. This method isolates highly motile sperm while filtering out debris and immotile cells. Studies show that microfluidics improve embryo quality, increase pregnancy rates, and may lead to higher euploidy rates. Additional benefits include improved safety, scalability, and shorter preparation times.

DETAILED DESCRIPTION:
In assisted reproductive technology (ART), the aim of sperm preparation is to select competent spermatozoa with the highest fertilization potential to be used for insemination by intracytoplasmic sperm injection (ICSI). This makes the process of selecting sperm highly important. Several methods have been developed to mimic some of the natural selection processes that exist in the female reproductive tract. Compared to the conventional sperm preparation techniques such as density gradient or sperm wash, microfluids can select sperm by controlling fluid dynamics within millimeter diameter capillaries in two parallel laminar flow channels, mimicking what potentially sperm experiment in the female genital tract without using centrifuge which can cause DNA sperm fragmentation. Hence, this technique could select spermatozoa with increased motility since motile spermatozoa can move through the flows and be eluted separately, while the debris and immotile cells are passively transported from the entrance to the exit of the capillary canal. There is scientific evidence that for couples undergoing ICSI, the spermatozoa that were selected by using microfluids resulted in a better-quality embryo which leaded to higher pregnancy outcomes. Also, literature suggest that euploidy rates of embryos obtained using microfluids are higher that using conventional sperm sample preparation. Among the advantages that microfluidics certainly offer are, safety, scalability and reduction sperm samples preparation times.

ELIGIBILITY:
Inclusion Criteria:

1. Women with at least 8 MII per cycle after denudation (AFC≥8).
2. Women of all ages.
3. All embryo qualities ≥BL3CC at the time of biopsy on day 5, 6 and/or 7.
4. Fresh sperm used from ejaculate with a concentration ≥1 mill/ml and ≥10% motility (A+B).
5. Sperm samples with a minimum of 2 ml.

Exclusion Criteria:

* Frozen oocytes samples with severe oligospermia (≤1mill/ml).
* PGT-M cases
* Sperm with > 1M/ml of round cells

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of sperm preparation time between microfluidic and gradient methods. | Immediately post-processing
  To evaluate and compare the time (in minutes) required to prepare sperm samples using microfluidic technology versus conventional density gradient centrifugation from the same ejaculate sample.
Comparison of euploidy rates in embryos derived from microfluidic versus gradient-prepared sperm. | Up to embryo biopsy (Day 5 or 6 post-fertilization)
  To compare the percentage of chromosomally normal (euploid) embryos, as determined by preimplantation genetic testing for aneuploidy (PGT-A), following fertilization using sperm processed via microfluidic versus gradient methods from the same semen sample.

SECONDARY OUTCOMES:
Comparison of post-processing semen parameters between microfluidic and gradient sperm preparation methods | Immediately post-processing
  To assess and compare motility (%) of sperm after preparation using microfluidic and gradient methods from the same sample.
Comparison of post-treatment semen parameters with pregnancy rates to evaluate the influence of sperm preparation methods on clinical outcomes. | From enrollment to the end of treatment at 1 year
  This objective aims to evaluate the correlation between post-treatment semen parameters-including sperm motility (%) measured by computer-assisted semen analysis (CASA), sperm concentration (million/mL) measured by manual counting using a Makler chamber, and morphology (% normal forms) assessed via strict criteria under microscopy-and clinical pregnancy rate (% of patients with confirmed intrauterine pregnancy by ultrasound). The comparison will be made between samples prepared using microfluidic and gradient sperm preparation methods. The goal is to determine whether higher values in semen quality parameters following preparation correlate with increased clinical pregnancy rates, providing quantifiable evidence of each technique's effectiveness in assisted reproductive treatments.
Comparison of fertilization rates between sperm processed via microfluidic and gradient methods | Day 1 post-insemination
  To evaluate the percentage of metaphase II oocytes successfully fertilized (2PN) using sperm prepared by each method.
Comparison of blastulation and utilization rates of embryos derived from microfluidic vs. gradient sperm preparation | Days 5-7 post-insemination
  To compare the percentage of embryos reaching the blastocyst stage (blastulation rate) and the percentage of usable blastocysts (utilization rate) between the two sperm preparation methods.
Number of Participants with Blastocyst Biopsy on Day 5, Day 6, or Day 7 by Sperm Preparation Method (Microfluidic vs. Gradient) | Day 5 to Day 7 post-insemination
  To determine whether the distribution of blastocyst biopsy days (Day 5 to Day 7 post-insemination) differs between the two sperm preparation methods.
Comparison of blastocyst morphological quality (expansion) between sperm preparation methods | Day 5-7 post-insemination
  Comparison of blastocyst expansion grade assessed immediately before biopsy using the modified Gardner scoring system.
  Scale: BL1-BL6 BL1: Blastocoel less than half of embryo volume (early blastocyst) BL2: Blastocoel at least half of embryo volume (early blastocyst) BL3: Full blastocyst, blastocoel completely fills embryo BL4: Expanded blastocyst with thin zona pellucida BL5: Herniation of cells through zona pellucida BL6: Blastocyst completely escaped from zona pellucida Interpretation: Higher scores indicate more advanced blastocyst development.
Mean Time to Key Embryo Developmental Milestones (2-Cell, 4-Cell, Blastocyst) by Sperm Preparation Method | From fertilization to blastocyst stage (Days 0-7)
  To compare mean time (in hours post-insemination) for embryos to reach the 2-cell, 4-cell, and blastocyst stages between microfluidic and gradient sperm preparation groups. All timepoints will be reported separately within the same outcome table. Unit of Measure: Hours.
Comparison of post-processing semen parameters between microfluidic and gradient sperm preparation methods | Immediately post-processing
  To assess and compare sperm concentration (million/mL) after preparation using microfluidic and gradient methods from the same sample.
Comparison of post-processing semen parameters between microfluidic and gradient sperm preparation methods | Immediately post-processing
  To assess and compare sperm morphology (% normal forms), after preparation using microfluidic and gradient methods from the same sample.
Comparison of post-processing semen parameters between microfluidic and gradient sperm preparation methods | Immediately post-processing
  To assess and compare sperm DNA fragmentation index (DFI, %) after preparation using microfluidic and gradient methods from the same sample.
Comparison of blastocyst morphological quality ( inner cell mass - ICM, ) between sperm preparation methods | Day 5-7 post-insemination
  Comparison of inner cell mass (ICM) quality using the modified Gardner scoring system, assessed immediately before biopsy.
  Scale: A-D A: Numerous tightly packed cells (best quality) B: Several loosely packed cells C: Very few cells D: No cells or >50% degenerated cells Interpretation: Grade A indicates the highest ICM quality.
Comparison of blastocyst trophectoderm quality (TE grades) between sperm preparation methods | Day 5-7 post-insemination
  Description: Comparison of trophectoderm (TE) quality using the modified Gardner scoring system, assessed immediately before biopsy.
  Scale: A-D A: Many cells forming a cohesive TE B: Several cells forming a loose epithelium C: Few cells with abnormal disposition D: Very few irregular, necrotic-appearing cells Interpretation: Grade A indicates the highest TE quality.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
as per request

REFERENCES:
- [Background] Chinnasamy T, Behr B, Demirci U. Microfuidic sperm sorting device for selection of functional human sperm for IUI application. Fertil Steril. 2016;105:e17-8. https://doi.org/10.1016/j.fertn stert.2015.12.063.
- [Background] Heydari A, Zabetian Targhi M, Halvaei I, Nosrati R. A novel microfluidic device with parallel channels for sperm separation using spermatozoa intrinsic behaviors. Sci Rep. 2023 Jan 21;13(1):1185. doi: 10.1038/s41598-023-28315-7. PMID 36681743
- [Background] Huang CH, Chen CH, Huang TK, Lu F, Jen Huang JY, Li BR. Design of a gradient-rheotaxis microfluidic chip for sorting of high-quality Sperm with progressive motility. iScience. 2023 Jul 17;26(8):107356. doi: 10.1016/j.isci.2023.107356. eCollection 2023 Aug 18. PMID 37559897
- [Background] Fang Y, Wu R, Lee JM, Chan LHM, Chan KYJ. Microfuidic invitro fertilization technologies: transforming the future of human reproduction. TrAC Trends Anal Chem. 2023;160:116959. https:// doi.org/10.1016/j.trac.2023.116959.
- [Background] Bastuba M, Cohen M, Bastuba A, Campbell P. Microfluidic sperm separation device dramatically lowers DFI. Fertil Steril. 2020;113(4, Supplement):E44 https://doi.org/10.1016/j.fertnstert.2020.02.096.
- [Background] Leung ETY, Lee CL, Tian X, Lam KKW, Li RHW, Ng EHY, Yeung WSB, Chiu PCN. Simulating nature in sperm selection for assisted reproduction. Nat Rev Urol. 2022 Jan;19(1):16-36. doi: 10.1038/s41585-021-00530-9. Epub 2021 Nov 5. PMID 34741158
- [Background] Quinn MM, Jalalian L, Ribeiro S, Ona K, Demirci U, Cedars MI, Rosen MP. Microfluidic sorting selects sperm for clinical use with reduced DNA damage compared to density gradient centrifugation with swim-up in split semen samples. Hum Reprod. 2018 Aug 1;33(8):1388-1393. doi: 10.1093/humrep/dey239. PMID 30007319
- [Background] Whitesides GM. The origins and the future of microfluidics. Nature. 2006 Jul 27;442(7101):368-73. doi: 10.1038/nature05058. PMID 16871203
- [Background] Vaughan DA, Sakkas D. Sperm selection methods in the 21st century. Biol Reprod. 2019 Dec 24;101(6):1076-1082. doi: 10.1093/biolre/ioz032. PMID 30801632
- [Background] ESHRE Guideline Group on Good Practice in IVF Labs; De los Santos MJ, Apter S, Coticchio G, Debrock S, Lundin K, Plancha CE, Prados F, Rienzi L, Verheyen G, Woodward B, Vermeulen N. Revised guidelines for good practice in IVF laboratories (2015). Hum Reprod. 2016 Apr;31(4):685-6. doi: 10.1093/humrep/dew016. Epub 2016 Feb 17. PMID 26908842
- [Background] Vander Borght M, Wyns C. Fertility and infertility: Definition and epidemiology. Clin Biochem. 2018 Dec;62:2-10. doi: 10.1016/j.clinbiochem.2018.03.012. Epub 2018 Mar 16. PMID 29555319
- [Background] CDC. 2016-National Summary Report-Assisted Reproductive Technology; US Department of Health. Human Service: Washington, DC, USA, 2018.
- [Background] De Munck N, El Khatib I, Abdala A, El-Damen A, Bayram A, Arnanz A, Melado L, Lawrenz B, Fatemi HM. Intracytoplasmic sperm injection is not superior to conventional IVF in couples with non-male factor infertility and preimplantation genetic testing for aneuploidies (PGT-A). Hum Reprod. 2020 Feb 29;35(2):317-327. doi: 10.1093/humrep/deaa002. PMID 32086522
- [Background] Lara-Cerrillo S, Raquel Jimenez Macedo A, Hortal O, Rosado Iglesias C, Lacruz Ruiz T, Carrera J, Garcia Peiro A. Impact of Microfluidic Sperm Sorting on Embryonic Euploidy in Infertile Patients with Sperm DNA Damage: A Retrospective Study. Int J Fertil Steril. 2024 Oct 30;18(4):417-423. doi: 10.22074/ijfs.2024.2007775.1499. PMID 39564835